CLINICAL TRIAL: NCT02492152
Title: Randomised ,Open Label in Meir Medical Center. Study the Potential of Dianatal Gel to Reduce the Rate of Episiotomy and Vaginal Tears in Birth
Brief Title: Does the Use of Dianatal Reduce the Rate of Episiotomy and Vaginal Tears in Birth?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Biron tal, MD, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0090-15
Record Dates: First submitted 2015-06-30; First posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Vaginal Tearing
Keywords: women; active labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Women who will not be using this medicine that is checked.
- Study group (Experimental): Women who will use DIANATAL according to manufacturer's protocol from the stage of active labor.
  Interventions: Device: Study group

INTERVENTIONS:
Device: Study group — Dianatal
  Arms: Study group

SUMMARY:
The purpose of the study is to see whether the use of DIANATAL during active labor, reduces the rates of episiotomy and vaginal tears.

DETAILED DESCRIPTION:
The risk for vaginal tears during birth is about 20%. These tears require surgical repair, are painful and make the recovery of the mother more difficult. Less commonly there is a risk of tear infection and regional scarring that make intercourse more difficult. Moreover, according to some studies, it appears that there is a link between damage to the pelvic floor and vagina during labor and Urinary incontinence in stress later in life.

It is clear that there is an advantage for the prevention of vaginal tears. Dianatal is a gel preparation, designed for use in births, in order to reduce the rate of vaginal tears and possibly shorten the second stage of labor.

Tested and found that using the gel reduces friction on tissue in processes simulating pressure of birth and therefore it is less likely to see tears in the vaginal tissue when using gel.

The product is approved for use by the ministry of health, was safety approved by regulatory bodies in Switzerland - the country of production.

So far, there is only one study published in the professional literature. The study found that using the gel at birth, reduces the duration of the second stage (full opening to the birth of the fetus) and reduces the rate of tears. The aim of the work was to investigate the effect of the product on the duration of labor. Women on their first birth, were divided randomly into two groups, one was treated with Dianatal from the stage of active labor, and the other group did not receive any treatment. In each research group were about ninety women. This is the single research in one population. In addition, the research group is too small to have statistical power in order to answer issues related to the number of vaginal tears and the need to perform episiotomies.

Considering such a significant issue for a woman who is giving birth and for the medical staff dealing with the newborn and in light of the minority research information on this subject, it is clear that there is room for further research.

Women who meet the inclusion criteria will be recruit to the research when arriving in the delivery room. They will sign the consent form and will be computerized randomized to one of two groups:

The study group - using DIANATAL according to manufacturer's protocol from their being in active labor.

The control group - women with the same conditions that will not be using this medicine that is checked.

The following data will be collected: medical background, pregnancy complications, preparations that were used to reduce the risk of birth tears before birth (perineal massage, EPINO), the duration of the stages in labor, use of epidural, neonatal weight, whether episiotomy or vaginal tears that required surgical intervention ( sewing) were done, post delivery process.

A comparison between the two groups will be made respectively with the results of the study that were defined.

ELIGIBILITY:
Inclusion Criteria:

Women on their first Childbirth

* Singleton pregnancy
* Over 37 weeks of pregnancy
* In active labor
* Women who intend to have a vaginally birth
* Women aged 18-45

Exclusion Criteria:

* Multiple pregnancy
* Births before 37 weeks
* History of tear degree III or more
* Women who intended to give birth by Caesarean section

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-04 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
number of women who will go through episiotomy and vaginal tears during birth | A year and a half

SECONDARY OUTCOMES:
Time of delivery | A year and a half
Number of women who will have post-delivery complications such as fever after childbirth, vaginal hematomas requiring intervention, long hospitalizations after birth. | A year and a half
Number of spontaneous vaginal births (that are not Instrumental deliveries) | A year and a half

REFERENCES:
- [Background] Eason E, Labrecque M, Wells G, Feldman P. Preventing perineal trauma during childbirth: a systematic review. Obstet Gynecol. 2000 Mar;95(3):464-71. doi: 10.1016/s0029-7844(99)00560-8. PMID 10711565
- [Background] Riener R, Leypold K, Brunschweiler A, Schaub A, Bleul U, Wolf P. Quantification of friction force reduction induced by obstetric gels. Med Biol Eng Comput. 2009 Jun;47(6):617-23. doi: 10.1007/s11517-009-0460-1. Epub 2009 Feb 24. PMID 19238473
- [Background] Schaub AF, Litschgi M, Hoesli I, Holzgreve W, Bleul U, Geissbuhler V. Obstetric gel shortens second stage of labor and prevents perineal trauma in nulliparous women: a randomized controlled trial on labor facilitation. J Perinat Med. 2008;36(2):129-35. doi: 10.1515/JPM.2008.024. PMID 18211256